CLINICAL TRIAL: NCT03897036
Title: A Phase I, Multi-Center, Open-Label, Treatment Duration Increment, Expansion, Safety, and Pharmacodynamic Study of CX-4945 Administered Orally Twice Daily to Patients With Advanced Basal Cell Carcinoma
Brief Title: Treatment Duration Increment and Pharmacodynamic Study of CX-4945 in Patients With Basal Cell Carcinoma (BCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Senhwa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CX-4945-07
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma, Basal Cell
Keywords: Advanced Basal Cell Carcinoma; laBCC; Locally Advanced Basal Cell Carcinoma; mBCC; Metastatic Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — silmitasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment-Duration-Increment (Experimental): CX-4945 capsules at 1000mg BID x 28 days/cycle
  Interventions: Drug: CX-4945
- Expansion (Experimental): CX-4945 capsules at 1000mg BID x 28 days/cycle
  Interventions: Drug: CX-4945

INTERVENTIONS:
Drug: CX-4945 — API powder-in-capsule in 200 mg strength

SUMMARY:
This study is to determine the recommended phase II dose (RP2D) and schedule of CX-4945 when administered orally twice daily for 28 consecutive days, in a 4-week (28 days) cycle, in patients with locally advanced or metastatic basal cell carcinoma (BCC). The safety and tolerability of CX-4945, preliminary evidence of antitumor effect, and the effect of CX-4945 treatment on the Hh signaling pathway will also be evaluated in this study.

DETAILED DESCRIPTION:
Basal cell carcinomas require the hedgehog (Hh) pathway for growth. Hh binding relieves the inhibitory effect of PTCH1 on Smoothened (SMO). Signal transduction by SMO then leads to the activation and nuclear localization of GLI1 transcription factors and induction of Hh target genes, many of which are involved in proliferation, survival, and angiogenesis. Hedgehog pathway inhibitors, such as vismodegib6 and sonidegib phosphate, target the G-protein-coupled receptor Smoothened (SMO) and are recommended as first-line treatment for advanced BCC or mBCC by the National Comprehensive Cancer Network. CK2 affects the terminal-most Hh signaling components. Given the roles of CK2 on the terminal step of the hedgehog signaling pathway, CK2 inhibition is unlikely to be overcome by downstream mutations within this pathway. These data thus suggest an immediately practical application of CX-4945 in Hh-driven tumors and possibly tumors resistant to SMO inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written IRB-approved informed consent.
2. Men and women age ≥ 18 years
3. ECOG Performance status 0 or 1
4. For patients with mBCC, histologic confirmation of distant BCC metastasis (e.g., lung, liver, lymph nodes, or bone), with metastatic disease that is RECIST measurable using CT or MRI

   Phase I Expansion:

   If a patient with locally advanced BCC also has a tumor that is not contiguous with cutaneous BCC, e.g., regional lymph nodes (if confirmed on biopsy as BCC and RECIST measurable), the patients should be considered as having mBCC and should be enrolled in the mBCC cohort
5. For patients with locally advanced BCC, histologically confirmed disease with at least one lesion that was 10 mm or more in at least 1 dimension by color photograph that is considered to be inoperable or medical contraindication to surgery (see below), in the opinion of a Mohs dermatologic surgeon, head and neck surgeon, or plastic surgeon
6. Acceptable medical contraindications to surgery include:

   1. BCC that has recurred in the same location after two or more surgical procedures and curative resection is deemed unlikely
   2. Anticipated substantial morbidity and/or deformity from surgery (e.g., removal of all or part of a facial structure, such as nose, ear, eyelid, eye; or requirement for limb amputation)
   3. Other conditions considered to be medically contraindicating must be discussed with the Medical Monitor before enrolling the patient.
7. For all patients, smoothened inhibitor must have been previously administered for their locally advanced or metastatic BCC, unless smoothened inhibitor is inappropriate (e.g., patient has received a smoothened inhibitor but became intolerant to the therapy). For patients whose BCC has been treated with smoothened inhibitor, disease must have progressed after treatment.
8. For patients with locally advanced BCC, radiotherapy must have been previously administered for their locally advanced BCC, unless radiotherapy is contraindicated or inappropriate (e.g., hypersensitivity to radiation due to genetic syndrome such as Gorlin syndrome, limitations because of location of tumor, or cumulative prior radiotherapy dose). For patients whose locally advanced BCC has been irradiated, disease must have progressed after radiation.
9. Previous Therapy

   * Surgery: Previous surgery is permitted provided that a minimum of 28 days (4 weeks) have elapsed between any major surgery and date of registration, and that wound healing has occurred.
   * Cytotoxic Chemotherapy: There is no limit to the number of prior regimens received.
   * Other Systemic Therapy: Previous treatment with Hh pathway antagonists is not allowed (except for Smoothened inhibitors). There is no limit to the other prior therapies received

   Patients must have recovered (to baseline or ≤ grade 1) from all reversible toxicity related to prior chemotherapy or systemic therapy and have adequate washout as follows:

   Longest of one of the following:
   * Two weeks,
   * 5 half-lives for investigational agents,

     * For anti-cancer therapies with half-lives > 8 days, a washout period of at least 28 days will be acceptable,
   * Standard cycle length of standard therapies.
10. Patients with nevoid BCC syndrome (Gorlin syndrome) may enroll in this study but must meet the criteria for locally advanced or metastatic disease listed above.
11. For patients with locally advanced BCC, willingness to consent to biopsy of tumor(s) at baseline and during the study, as mandated by the protocol
12. Adequate hematopoietic capacity, as defined by the following:

    * Hemoglobin ≥ 9.0 g/dL and not transfusion dependent
    * Platelets ≥ 100,000/mm3
    * Absolute neutrophil count ≥ 1500 cells/mm3
13. Adequate hepatic function, as defined by the following:

    * AST and ALT ≤ 2.5 times upper limit of normal (ULN) or ≤ 5 times ULN if liver metastases are present
    * Total bilirubin ≤ 1.5 x ULN or within 3x the ULN for patients with Gilbert disease
    * Albumin ≥ 3.0 g/dL
14. Adequate renal function, as defined by the following:

    * Renal: calculated creatinine clearance >45 mL/min for patients with abnormal, increased, creatinine levels (Cockcroft-Gault formula).
15. Women/men of childbearing potential must have agreed to use two effective contraceptive methods while on study and for 6 months after the last dose of CX-4945 (see Appendix D for definition of women of childbearing potential and acceptable and unacceptable methods of contraception)

Exclusion Criteria:

1. Tumor histology consistent with basosquamous carcinoma (basal cell carcinoma with squamous differentiation or metatypical carcinoma).
2. Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a man father a child, or a woman become pregnant or suspect she is pregnant while participating in this study, he or she should inform the treating physician immediately.
3. Concurrent non-protocol-specified anti-tumor therapy (e.g., chemotherapy, other targeted therapy, radiation therapy, or photodynamic therapy)

   * For patients with multiple cutaneous BCCs at baseline that are not designated by the investigator as target lesions, treatment of these non-target BCCs with surgery may be permitted but must be discussed with the Medical Monitor prior to any surgical procedure.
   * For patients with locally advanced BCC whose target lesion(s) is/are inoperable at baseline but is/are later deemed potentially operable because of tumor response to CX-4945, surgery with curative intent may be permitted but must be discussed with the Medical Monitor prior to any surgical procedure.
4. History of other malignancies within 3 years of Day 1, except for tumors with a negligible risk for metastasis or death, such as adequately treated squamous-cell carcinoma of the skin, ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix
5. Active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
6. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk from treatment complications
7. Difficulty with swallowing oral medications
8. Chronic diarrhea (excess of 2-3 stools/day above normal frequency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Huang, MD, Study Director — Senhwa Biosciences
Locations (6):
- United States (6):
  - HonorHealth Research & Innovation Institute, Scottsdale, Arizona
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Texas Oncology, P.A., Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled on April 16, 2019. Last subject visit occurred on January 25, 2024.
  Six investigators at different study centers in the United States each enrolled at least one subject.
  A total of 3 to 6 subjects were to be enrolled to define the RP2D, and 20 subjects were planned to be enrolled in the expansion part of the study. A total of 25 subjects were enrolled: 8 subjects in Cohort 1 and 17 subjects in Cohort 2.
Pre-assignment Details: Of 30 screened subjects, 25 met all inclusion/exclusion criteria and were enrolled into the study.
Groups:
- Treatment-Duration-Increment; Expansion: 1000 mg BID × 28 days/cycle
  CX-4945: API powder-in-capsule in 200 mg strength
Period: Overall Study
Arm/Group | Treatment-Duration-Increment | Expansion
Started | 8 | 17
Completed (There was only one DLT at the 1000mg BID x28 day/ cycle dosing schedule. In compliance with the design of the protocol, this dosing schedule of 1000mg BID x28 day/ cycle was determined to be the RP2D, and Expansion cohort was opened using the same dosing schedule.) | 8 | 16
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-Duration-Increment | Expansion | Total
Number analyzed (Participants) | 8 | 17 | 25
Age, Continuous [Median (Full Range); unit: years] | 65 [40 to 81] | 64 [37 to 83] | 64 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 5 | 12 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 17 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 17 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 17 | 25

OUTCOME MEASURES:

1. Primary Outcome: Determination of RP2D
Description: Determination of RP2D for the expansion cohorts
Time Frame: Cycle 1, twenty-eight (28) day continuous dosing schedule
Measure: Number; unit: mg
Arm/Group | Treatment-Duration-Increment
Number analyzed (Participants) | 8
mg | 1000

ADVERSE EVENTS:
Time Frame: Adverse events data were collected After informed consent, but prior to initiation of study drug, only SAEs caused by a protocol-mandated intervention will be collected (e.g., SAEs related to invasive procedures such as biopsies, medication washout, or no treatment run-in). After initiation of study drug, all AEs and SAEs regardless of attribution will be collected until 30 days following the last administration of study treatment or study discontinuation/termination, whichever is later.
Arm/Group | Treatment-Duration-Increment | Expansion
All-Cause Mortality (participants affected / at risk) | 0/8 | 1/17
Serious Adverse Events (participants affected / at risk) | 2/8 | 3/17
Other Adverse Events (participants affected / at risk) | 8/8 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Duration-Increment (N=8) | Expansion (N=17)
COVID-19 (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Superventricular Tachycardia (Cardiac disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Duration-Increment (N=8) | Expansion (N=17)
Diarrhoea (Gastrointestinal disorders) | 8 | 14
Nausea (Gastrointestinal disorders) | 5 | 9
Vomiting (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 4
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal irritation (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 4
Lymphocyte count decreased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Blood bicarbonate increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 0 | 2
Lymphocyte count increased (Investigations) | 0 | 1
Fatigue (General disorders) | 2 | 2
Asthenia (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No submission for publication or public disclosure by Institution or Investigator will be made until after publication of the multicenter results. After the first to occur of (i) publication of the multicenter results, (ii) notification by Sponsor that such a multicenter submission is no longer planned, or (iii) eighteen months after the Completion Date of the Study as defined in 42 CFR 11.10, Institution and Investigator may publish or publicly present the Study Data.

DOCUMENTS (2):
  • Study Protocol (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT03897036/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03897036/SAP_001.pdf